CLINICAL TRIAL: NCT03954678
Title: Prospective Randomized Study of Exercise in Patients Undergoing Urologic Surgery
Brief Title: Exercise in Patients Undergoing Urologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: vmaster (Unknown)
Responsible Party: Principal Investigator, Kenneth Ogan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00044694
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Complication
Keywords: Exercise; Nutrition supplement; Surgery
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants randomized to the activity intervention will aim for taking 10,000 steps per day and completing strength training exercises three times per week.
  Interventions: Behavioral: Exercise Group
- Nutrition Group (Active Comparator): Participants randomized to the nutrition intervention will consume a liquid over-the-counter nutrition supplement two times per day.
  Interventions: Dietary Supplement: Nutrition Group

INTERVENTIONS:
Behavioral: Exercise Group — For the first two days after their pre-operative visit, participants will be asked to continue their present level of exercise and activity, which will be monitored by pedometer. Participants will begin the activity intervention on study Day 3. Participants will be instructed to take 10,000 steps per day, recording their daily steps with a pedometer. Participants also will be provided with resistance bands and instructed on how to safely perform 10 whole-body strength training exercises. They will be instructed to perform the exercises once per day, three days a week. Participants will complete the exercise intervention until they have surgery, which is typically 12 to 48 days after the pre-operative visit.
  Arms: Exercise Group
Dietary Supplement: Nutrition Group — Participants in the nutrition group will be provided with a liquid over-the-counter nutrition supplement (i.e. Boost or Ensure) to consume. Participants will be instructed to consume 1 bottle, 2 times per day, beginning 5 days before surgery and continuing 5 days post-operatively.
  Arms: Nutrition Group

SUMMARY:
Patients who are being scheduled for an operative procedure with an inpatient postoperative stay are eligible for this study. Participants will be selected to start a physical fitness plan or a nutrition plan at the time of surgical scheduling. Each participant will be asked to continue their current lifestyle for two days after their pre-operative appointment to get a baseline of activity (by pedometer and functional tests) and nutritional risk (by questionnaire). After two days, patients in the activity group will start their activity plans. They will be encouraged to get 10,000 steps per day and to perform whole body strength training exercises 3 times a week. Five days before and after surgery, participants in the nutrition group will be asked to consume a standard liquid nutrition supplement (i.e. Boost or Ensure) two times per day. Participants in the activity group will record steps and number of strength training sessions completed, while patients in the nutrition group will record the number of supplements consumed.

DETAILED DESCRIPTION:
Increases in physical activity and nutritional status are associated with improvements in a number of health conditions, including coronary artery disease, hypertension, stroke, insulin sensitivity, osteoporosis, and depression. Regretfully, despite the evidence supporting the benefits of physical activity, greater than half of adults in the United States do not get adequate activity and approximately one quarter do not get any activity. As such, many people, especially the elderly and those with comorbid diseases, have low levels of physical fitness. Additionally, up to 45% of community dwelling older adults are malnourished. Patients undergoing surgery with poor exercise tolerance and suboptimal nutritional status may be at an increased risk of perioperative complications. Thus, increasing physical activity and dietary intake quality prior to surgery is recommended, to hopefully decrease these risks. The primary objective is to determine if recommended physical activity or dietary intake results in an increase in patient physical function performance and if so, to what extent. The secondary goal is to examine if increased exercise or nutrition reduces perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for operative procedure with an inpatient postoperative stay are eligible for this study
* Patients willing and able to give blood sample as part of standard of care labs
* Patients willing and able to fill out questionnaire
* Patients who will fill out the step log daily
* Patients willing and able to sign informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  Body Mass Index is a weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters (kg/m^2) and used as an indicator of underweight, normal, overweight and obese weights.
Change in Standing Task Time | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  Participants will be timed, in seconds, to see how quickly they can stand up and sit down in a chair 5 times.
Change in 6 Minute Walk Test (6MWT) Distance | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  The 6 minute walk test (6MWT) assesses distance, in meters, walked over 6 minutes as a sub-maximal test of aerobic capacity and endurance.
Change in grip strength | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  Hand grip is measured in pounds using a dynamometer to test the maximum isometric strength of the hand and forearm muscles. Grip strength is a measurement of muscle strength and tends to decline with frail states.
Change in Timed Up and Go (TUG) Task | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  Participants will be timed, in seconds, to see how quickly they can rise from a chair, walk 3 meters, turn around, walk back, and sit down.
Change in Short-Length Food Frequency Questionnaire | Baseline, Day of surgery (up to 50 days after Baseline), Follow-up (30 days after surgery)
  Nutritional risk will be assessed with the Short-Length Food Frequency Questionnaire. This 18-item instrument asks participants how frequently they consume certain foods, such as alcohol, produce, grains, and fried foods. There is not a summary score for this questionnaire, rather, the researchers can examine changes over time in foods consumed in a variety of ways.

SECONDARY OUTCOMES:
Perioperative Complications | 30 days after surgery
  The number of perioperative complications will be compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No